CLINICAL TRIAL: NCT05580614
Title: Pairing tVNS and Exposure and Response Prevention to Improve Symptoms of OCD
Brief Title: Paired tVNS With ERP in OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: International OCD Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202101733; OCR41263 (Other: UF OnCore)
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: OCD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tVNS paired with 12 sessions of ERP (Active Comparator)
  Interventions: Device: tVNS
- Sham tVNS paired with 12 sessions of ERP (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Sham — MRI (Magnetic Resonance Imaging) paired ERP/Sham YBOCs(Yale-Brown Obsessive Compulsive Scale) (4,8,12) OCI-R (every other session). YBOCs and OCI-R will also be administered at intake and 4 weeks post treatment.
  Arms: Sham tVNS paired with 12 sessions of ERP
Device: tVNS — MRI (Magnetic Resonance Imaging) paired ERP/tVNS YBOC's (Yale-Brown Obsessive Compulsive Scale) (4, 8, 12) OCI-R (every other session). YBOCs and OCI-R will also be administered at intake and 4 weeks post treatment.
  Arms: Active tVNS paired with 12 sessions of ERP

SUMMARY:
In the proposed investigation, the investigator will develop pilot data for the use of tVNS (transcutaneous vagal nerve stimulation) to enhance efficacy of exposure and response prevention therapy (ERP) to improve treatment success in patients with OCD. This data will include tolerability information from therapists and patients with OCD, effect sizes on real world clinical outcomes for the combinatory treatment, and mechanistic data on brain changes associated with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 55
* Meet DSM-5 criteria for OCD, based on a structured clinical interview and who have a YBOCS score of 15 or higher, indicating at least moderate OCD severity
* Participants must be willing and able to provide informed consent.

Exclusion Criteria:

* Participants with major neurological conditions, autism spectrum disorder, psychosis, major uncorrected sensory deficit, and severe medical disease that may be associated with neurological effects.
* People with an active eating disorder that requires treatment, but we will not exclude people who are in remission.
* Current illicit or prescription drug abuse
* Participants who are receiving pharmacotherapy for their OCD or for other psychiatric disorders will not be excluded
* No medication changes will be allowed during the study, and participants must be on stable doses of medications for at least 6 weeks prior to entering the study. Prior ERP treatment (at least 12 months removed) is acceptable

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive-Compulsive Scale (Y-BOCS) | Baseline up to 1 month post treatment
  A test to rate the severity of obsessive-compulsive disorder (OCD) symptoms. The 10 Y-BOCS items are each scored on a four-point scale from 0 = "no symptoms" to 4 = "extreme symptoms." The sum of the first five items is a severity index for obsessions, and the sum of the last five an index for compulsions. Total scores on the measure range from 0 to 40, with a score of 0-7 indicating subclinical symptoms, 8-15 mild symptoms, 16-23 moderate symptoms, 24-31 severe symptoms and 32-40 extreme symptoms. The scale can also provide a subscale score for obsessions and compulsions (range 0-20) separately.

CONTACTS AND LOCATIONS:
Overall Officials: John Williamson, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No